CLINICAL TRIAL: NCT06030635
Title: Non-invasive Monitoring of Patients At Risk of Acute Compartment Syndrome (ACS) with CPMX1
Brief Title: ACS Monitoring Charité Berlin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Compremium AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1056
Record Dates: First submitted 2023-09-01; First posted 2023-09-11 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Compartment Syndromes
MeSH Terms: conditions — Compartment Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CPMX1 (Experimental): Compartment compressibility measurement using the CPMX1 device
  Interventions: Device: Measurement of compartment compressibility using the CPMX1 device

INTERVENTIONS:
Device: Measurement of compartment compressibility using the CPMX1 device — Patients will be monitored about every hour (+/- 30 min) for a total of 8 hours. Measurement time might be extended in case the patient undergoes trauma-related surgery during the measurement period and/or in case measurements are spaced further apart. Remaining measurements will be completed after the surgery. At each time point, three measurements of compartment compressibility will be conducted using the CMPX1 on both the affected (potential ACS) and healthy limb.

SUMMARY:
Compartment syndrome is a very serious musculoskeletal disorder, which can lead to devastating consequences, such as limb amputation and life-threatening conditions. It is a well described medical condition considered to be an orthopaedic emergency affecting all ages.

In the diagnosis of acute compartment syndrome, clinical suspicion supplemented by careful, repeated clinical examination continues to be the clinician's greatest tool. The classic signs and symptoms of acute compartment pressure are often listed as the 5 or 6 "Ps": Pain, Pressure, Pulselessness, Paralysis, Paresthesia, and Pallor. The diagnosis is typically not made by using equipment and it is difficult in the awake and oriented patient, becoming even more problematic in the polytrauma patient.

An alternative diagnostic method for compartment syndrome is invasive intra-compartmental pressure measurement via insertion of a pressure monitoring device into the muscle compartment. However, literature shows that commercially available intra compartmental pressure monitors have a highly variable intra-observer reproducibility and that user errors are common.

Compared to the invasive modalities or just experience of the surgeon, the CPMX1 shows promising advantages for the clinical application. Not only is the technology used for the CPMX1 device safe and non-invasive for the patient with only initial training required for the healthcare professionals, but it has also demonstrated high intra- and inter-observer reproducibility (as per bench tests and confirmed in clinical setting). Recently, two clinical studies ("SWISS_EVIDENCE" and "SWISS_CLEARANCE") were conducted using the CPMX1 in healthy volunteers in a real-world clinical environment. Results of these studies confirmed that the application of the CMPX1 in patient care is safe and validated the reliability of compressibility ratio measurement with the CPMX1 in healthy volunteers.

The use of the CPMX1 device therefore facilitates the measurements, as it is based on pre- existing ultrasound methods, and avoids any further risks to the patients compared to invasive compartmental pressure diagnosis methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to give consent
* Informed consent documented by signature
* Potential acute compartment syndrome (ACS) of the extremities (excl. hands, feet)
* Male or female
* Age 18 to 95 years
* Intact skin at the measurement site
* Open fracture up to Grade I if not in the measurement area

Exclusion Criteria:

* Potential Acute Compartment Syndrome (ACS) of both extremities considered
* Limb anomalies that could hinder the measurement
* Individuals who are deprived of liberty pursuant to an administrative order or court order or approval.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
Lowest CP Values [percent] (highest compartmental pressure) | During the procedure which will last 8 hours/patient (measurement time might be extended in case of trauma-related surgery during the measurement period and/or in case measurements are spaced further apart)
  Lowest CP Values [percent] (highest compartmental pressure) will be assessed from the difference in CP Values [percent] using the CPMX1 for a compartment at risk of ACS and compartment not at risk of ACS at the same time, contrasted by a pairwise t-test.

SECONDARY OUTCOMES:
CP Value [percent] trend over time | During the procedure which will last 8 hours/patient (measurement time might be extended in case of trauma-related surgery during the measurement period and/or in case measurements are spaced further apart)
  Each study patient will be monitored every hour for a total of 8 hours (measurement time might be extended in case of trauma-related surgery during the measurement period and/or in case measurements are spaced further apart) with the investigational device. The CP Value [percent] trend over time will be visualized per patient through plots.
CP Values [percent] from the compartments at risk of ACS and CP Values [percent] of compartment not at risk at the same time. | During the procedure which will last 8 hours/patient (measurement time might be extended in case of trauma-related surgery during the measurement period and/or in case measurements are spaced further apart)
  CP Value [percent] of extremities at risk and not at risk of ACS will be contrasted by a pairwise t-test.
Quotient CP Value [percent] | During the procedure which will last 8 hours/patient (measurement time might be extended in case of trauma-related surgery during the measurement period and/or in case measurements are spaced further apart)
  Quotient calculation will be performed between CP Value of affected and non-affected limb's compartment. Values will be contrasted between the groups.
Time of the lowest CP Values [percent] (highest compartmental pressure) for the compartment at risk of ACS | During the procedure which will last 8 hours/patient (measurement time might be extended in case of trauma-related surgery during the measurement period and/or in case measurements are spaced further apart)
  The mean time point for lowest CP Values [percent] and range will be calculated.
Usability and workflow assessment | At the end of the participation of each investigator to the clinical study (up to 5 months)
  Usability and workflow assessment will be evaluated through a practitioner's questionnaire which will be filled by each investigator at the end of the participation in the clinical investigation. The questionnaire will cover different aspects regarding usability and safety of the CPMX1 device.

OTHER OUTCOMES:
Assessment of adverse events | During the procedure which will last 8 hours/patient (measurement time might be extended in case of trauma-related surgery during the measurement period and/or in case measurements are spaced further apart)
  Safety of the device will be assessed by systematically reporting adverse events and serious adverse events (description, severity, relation to the procedure) and by monitoring the frequency and incidence of these events.
Assessment of device deficiencies | During the procedure which will last 8 hours/patient (measurement time might be extended in case of trauma-related surgery during the measurement period and/or in case measurements are spaced further apart)
  Safety of the device will be assessed by systematically reporting device deficiencies (description of the deficiency) and by monitoring the frequency and incidence of these events
New risk identification | At the end of the participation of each investigator to the clinical study (up to 5 months)
  The practitioner will be asked to identify any new risks arising when using the investigational device.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Gehlen, Dr med, Principal Investigator — Centrum für Muskuloskeletale Chirurgie Charité - Universitätmedizin Berlin
Locations (1):
- Centrum für Muskuloskeletale Chirurgie Charité - Universitätmedizin Berlin, Berlin, Germany, Germany

IPD SHARING:
Plan to Share IPD: No